CLINICAL TRIAL: NCT03366974
Title: Assessment of Change in CYP3A Activity by Route of Administration Using Metabolic Markers in Healthy Male Volunteers
Acronym: CYP_IVPO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Joo-Youn Cho, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CYP_IVPO
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Midazolam; Clarithromycin

STUDY DESIGN:
Intervention Model Description: An open-label, one-sequence, three-period study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CYP inhibition + IV/PO midazolam (Experimental): Period 1: Administration of Midazolam (IV) on day 1, Co-administration of Midazolam (IV) and Grapefruit juice on day 2
  Period 2: Administration of Midazolam (PO) on day 8, Co-administration of Midazolam (PO) and Grapefruit juice on day 9
  Period 3: Self-administration of Clarithromycin (PO) bid regimen on day 12-14, Co-administration of Midazolam (IV) and Clarithromycin (PO) on day 15, Co-administration of Midazolam (PO) and Clarithromycin (PO) on day 16
  Interventions: Drug: Midazolam; Drug: Clarithromycin; Dietary Supplement: Grapefruit juice

INTERVENTIONS:
Drug: Midazolam — Midazolam 5 mg PO, Midazolam 1 mg IV
Drug: Clarithromycin — Clarithromycin 500 mg bid
Dietary Supplement: Grapefruit juice — Grapefruit juice 500 mL

SUMMARY:
The study objective is to evaluate and validate of endogenous markers for the assessment of change in CYP3A activity by route of administration in Korean healthy subjects using metabolomics. In addition, we aim to screen novel endogenous marker, which could determine the total or intestinal CYP activity.

DETAILED DESCRIPTION:
This study is an open-label, one-sequence, three-period study. A total of 16 healthy male subjects will be enrolled. In period 1, subjects will be administered midazolam IV 1 mg, and co-administration of midazolam IV 1mg and grapefruit juice 500 mL. In period 2, subjects will be administered midazolam PO 5 mg, and co-administration of midazolam PO 5mg and grapefruit juice 500 mL. In period 3, subjects will be administered clarithromycin 500 mg for 3-days in b.i.d regimen prior to admission. Subjects will be administered midazolam IV 1mg and PO 5mg after admission.

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 19 to 50 years of age
* Weight: Within 17 - 28 of Body Mass Index (BMI)
* Subject who are reliable and willing to make themselves available during the study period, and subject who are willing to follow the study protocol, and give their written informed consent voluntarily.

Exclusion Criteria:

* History of hypersensitive reaction to medication (midazolam, aspirin, NSAID, antibiotics, benzodiazepine, erythromycin, macrolide)
* History of significant clinical illness needs medical caution, including cardiovascular, immunologic, hematologic, neuropsychiatric, respiratory, gastrointestinal, hepatic, or renal disease or other chronic disease history or evidence of drug abuse
* Subjects with evidence or a history of gastrointestinal disease (e.g, gastritis, Chron's disease) or with history of gastrointestinal surgery (except simple appendectomy or herniorrhaphy) that may affect assessment of PK characteristics of study drug
* Any of the following ECG abnormalities: QTcF > 450 msec
* History of apnea
* Subjects with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Subject whose systolic blood pressure is over 150 mmHg or below 90 mmHg and diastolic blood pressure is over 100 mmHg or below 50 mmHg
* Subjects with a history of drug abuse or a positive urine screening for drug abuse
* Subjects who have participated in any other clinical trial within three months prior to study drug administration
* Use any prescriptive medication, Korean traditional medication not considered acceptable by the clinical investigator during the last 14 days period before first dosing, or use any medication not considered acceptable by the clinical investigator during the last 7 days period before first dosing (if used medication is considered acceptable by investigator, patients can be included)
* Subjects who have donated a unit of whole blood within two months or blood components within one month prior to study drug administration
* Subjects who consume more than 21 units of alcohol per week (1 unit = 10 g of pure alcohol) or who are unable to abstain from drinking during the admission period
* Smokers (except for those who had quit for at least three months before the first administration of the IP)
* Subjects who consume or are unable to abstain from products containing grapefruit during study period
* Subjects who consume or are unable to abstain from products containing caffeine during study period
* Subjects who are positive for Hepatitis B, Hepatitis C, and HIV
* Subject who judged not eligible for study participation by investigator

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve of midazolam (AUClast) | Up to 12 hours after midazolam administration
  Pharmacokinetics of midazolam
Metabolic ratio of steroids | Up to 12 hours before/after midazolam administration
  endogenous metabolite profiles such as steroid (6beta-hydroxy-cortisol/cortisol, 6beta-hydroxy-cortisone/cortisone)
Clearance (CL) of midazolam | Up to 12 hours after midazolam administration
  Pharmacokinetics of midazolam

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Youn Cho, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea